CLINICAL TRIAL: NCT02783040
Title: A Study to Investigate the Effects of Multiple Doses of BI 425809 on the Single Dose Pharmacokinetics of Cytochrome P450 Substrates (Midazolam, Warfarin and Omeprazole) and a P Glycoprotein Substrate (Digoxin) Administered Orally in an Open-label, One-sequence Trial in Healthy Male Subjects
Brief Title: Interaction of BI 425809 With Midazolam, Warfarin, Omeprazole and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346.22; 2015-001371-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2016-03-23; First posted 2016-05-26 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Warfarin; Omeprazole; Digoxin; BI 425809

ARMS (4):
- single dose cocktail (Midazolam, Warfarin, Omeprazole) (Experimental)
  Interventions: Drug: Midazolam; Drug: Warfarin; Drug: Omeprazole
- single dose Midazolam (Experimental)
  Interventions: Drug: Midazolam
- single dose Digoxin (Experimental)
  Interventions: Drug: Digoxin
- multiple dose BI 425809 (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: Midazolam
  Arms: single dose cocktail (Midazolam, Warfarin, Omeprazole)
Drug: Warfarin
  Arms: single dose cocktail (Midazolam, Warfarin, Omeprazole)
Drug: Omeprazole
  Arms: single dose cocktail (Midazolam, Warfarin, Omeprazole)
Drug: Midazolam
  Arms: single dose Midazolam
Drug: Digoxin
  Arms: single dose Digoxin
Drug: BI 425809
  Other Names: Iclepertin
  Arms: multiple dose BI 425809

SUMMARY:
To assess the influence of multiple doses of BI 425809 on single dose pharmacokinetics of midazolam (CYP3A4 probe drug), warfarin (CYP2C9 probe drug), omeprazole (CYP2C19 probe drug) and digoxin (P-gp probe drug)

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), puls rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation
* Ready and able to use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the subject information

Exclusion criteria:

* Any finding in the medical examination (including blood pressure (BP), puls rate (PR) or electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | 0-119 hours
Cmax (maximum measured concentration of the analyte in plasma) | 0-119 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.22.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Desch M, Schlecker C, Hohl K, Liesenfeld KH, Chan T, Muller F, Wunderlich G, Keller S, Ishiguro N, Wind S. Pharmacokinetic-Interactions of BI 425809, a Novel Glycine Transporter 1 Inhibitor, With Cytochrome P450 and P-Glycoprotein Substrates: Findings From In Vitro Analyses and an Open-Label, Single-Sequence Phase I Study. J Clin Psychopharmacol. 2023 Mar-Apr 01;43(2):113-121. doi: 10.1097/JCP.0000000000001656. Epub 2023 Jan 26. PMID 36700734